CLINICAL TRIAL: NCT02273440
Title: The Effects of Multiple Doses of BIIL 284 BS on the Pharmacokinetics of a Single Dose of Theophylline in Healthy Male Volunteers (a Randomized, Double-blind, Placebo-controlled, Two-period, Two-way Crossover Study)
Brief Title: Effect of BIIL 284 BS on the Pharmacokinetics of Theophylline in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 543.7
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — amelubant; Theophylline

ARMS (2):
- BIIL 284 BS with theophylline (Experimental)
  Interventions: Drug: BIIL 284 BS; Drug: Theophylline
- Placebo with theophylline (Placebo Comparator)
  Interventions: Drug: Theophylline; Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS
  Arms: BIIL 284 BS with theophylline
Drug: Theophylline
Drug: Placebo
  Arms: Placebo with theophylline

SUMMARY:
To evaluate the effect of multiple doses of BIIL 284 BS on the pharmacokinetics of a single dose of theophylline.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated prior to participation into the study (including medication washout)
* All volunteers in the study should be healthy males, aged 18-50 years (inclusive) and willing to use condoms until 60 days after the last dose
* All volunteers should be within +- 20% of their ideal body weight (Metropolitan Scale, 1983)
* Non-smokers (volunteers who have never smoked) or ex-smokers for at least one year with a smoking history, no greater than five pack-years (1 pack year = 20 cigarettes per day for one year)
* Ability to comply with the concomitant therapy restrictions
* Volunteers will be off all prescription drugs. O.T.C. drugs must be discontinued for at least two weeks prior to the first dose of study drug. If throughout the study, volunteers need any O.T.C. medication, the investigator will call the clinical monitor and this will be reviewed on a case-by-case bases. Restrictions for different medications apply
* Volunteers will have no evidence of a clinically relevant concomitant disease based upon complete medical history, physician global assessment, complete physical examination, ECG, and clinical laboratory tests

Exclusion Criteria:

* Viral respiratory tract infection, respiratory tract infection within the six weeks preceding the first day of dosing with study medication
* Small of difficult to locate arm or hand veins that would impair the clinician's ability to draw blood samples or to place a venous catheter
* Volunteers with a known drug or alcohol dependence (presence of dependency for 10 years) or who drink more than 60 g of alcohol per day
* History of significant allergic reactions to drugs or sensitivity to aspirin or positive drug screen
* Use of an investigational new drug in the preceding 3 months or six half-lives (whichever is greater) prior to the first screen at Visit 1
* Donation of blood during the preceding 3 months of Visit 1
* Volunteers receiving hyposensitization therapy whom are not on a stable dose for the last three months before Visit 1
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Volunteers with disease of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/hypersensitivity (including drug allergy) with is deemed relevant to the trial as judged by the investigator
* Volunteers with eosinophilia > 7%
* Volunteers who received any other drugs which might influence the results of the trial during the week previous to the start of the study
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2000-05; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Plasma levels of theophylline | up to 72 hours after theophylline administration
Area under the curve from zero extrapolated to infinity (AUC0-infinity) | up to 72 hours after theophylline administration
Peak plasma concentration (Cmax) for theophylline | up to 72 hours after theophylline administration

SECONDARY OUTCOMES:
Time to peak plasma concentration (tmax) | up to 72 hours after theophylline administration
Terminal half-life (t1/2) | up to 72 hours after theophylline administration
Total mean residence time (MRTtot) | up to 72 hours after theophylline administration
Total clearance after oral administration (CLtot/F) | up to 72 hours after theophylline administration
Volume of distribution during terminal phase after oral administration (Vz/F) | up to 72 hours after theophylline administration
Area under the concentration time curve at steady state (AUC,ss) for BIIL 315 ZW | up to 72 hours after theophylline administration
Peak plasma concentration at steady state (Cmax,ss) for BIIL 315 ZW | up to 72 hours after theophylline administration
Number of patients with adverse events | up to 5 days after last theophylline administration
Number of patients with clinically significant findings in vital signs | up to 3 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 3 days after last drug administration
Number of patients with clinically significant findings in 12-lead ECG | up to 3 days after last drug administration